CLINICAL TRIAL: NCT06445764
Title: Enhancing Trauma Cardiopulmonary Resuscitation Simulation Training With the Use of Virtual Reality (Trauma SimVR): Protocol for a Randomized Controlled Trial
Brief Title: Traumatic Cardiac Arrest and Trauma SimVR Training
Acronym: Trauma SimVR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical problems with VR scenario development
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Josef Michael Lintschinger, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1388/2023
Record Dates: First submitted 2024-05-26; First posted 2024-06-06 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-07

CONDITIONS: Virtual Reality; Heart Arrest
Keywords: in-hospital cardiac arrest; Education, Medical
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- e-learning (Other)
  Interventions: Other: e-learning
- Virtual reality training (Other)
  Interventions: Other: Virtual reality training

INTERVENTIONS:
Other: e-learning — Participants will complete an e-learning course over a two-week period that focuses on skills and knowledge related to the management of in-hospital cardiac arrest. This course prepares participants for an in-person assessment.
  Arms: e-learning
Other: Virtual reality training — Participants will complete a virtual reality training over a two-week period that focuses on skills and knowledge related to the management of in-hospital cardiac arrest. This training prepares participants for an in-person assessment.
  Arms: Virtual reality training

SUMMARY:
The goal of this single-center, prospective, randomized, controlled trial is to evaluate the effectiveness of using virtual reality technology to provide learners with skills and knowledge in the management of traumatic cardiac arrest in first-year residents at the emergency department.

The main question it aims to answer is:

Does the use of virtual reality in the context of trauma cardiopulmonary resuscitation training result in shorter times to order/perform pre-defined critical actions?

Participants will learn management skills for in-hospital traumatic cardiac arrest using either newly developed virtual reality software or e-learning focused on the same content.

ELIGIBILITY:
Inclusion Criteria:

* first-year residents at the emergency department
* only people who do not need eyeglasses for using VR

Exclusion Criteria:

- pre-disposition for cybersickness (motion sickness, pregnancy, pre-existing cybersickness)

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to critical action | evaluation within 4 weeks after study completion
  Expert-based assessment of the difference in time (seconds) to the predefined primary critical action between randomized groups in video recordings of an in-person assessment simulation.

SECONDARY OUTCOMES:
Time to secondary critical action #1 | evaluation within 4 weeks after study completion
  Expert-based assessment of the difference in time (seconds) to the predefined secondary critical action #1 between randomized groups in video recordings of an in-person assessment simulation.
Time to secondary critical action #2 | evaluation within 4 weeks after study completion
  Expert-based assessment of the difference in time (seconds) to the predefined secondary critical action #2 between randomized groups in video recordings of an in-person assessment simulation.
Number of unrecognized causes of traumatic cardiac arrest | evaluation within 4 weeks after study completion
  Expert-based assessment of the difference in unrecognized underlying causes of traumatic cardiac arrest between randomized groups in video recordings of an in-person assessment simulation.
Number of patients declared dead prematurely | evaluation within 4 weeks after study completion
  Expert-based assessment of the difference in the number of patients declared dead prematurely between the randomized groups in video recordings of an in-person assessment simulation.
Number of protocol deviations | evaluation within 4 weeks after study completion
  Expert-based assessment of the difference in the frequency of protocol deviations between randomized groups in video recordings of an in-person assessment simulation. Protocol deviations are listed in the study protocol and reflect the recommendations of the guidelines on which the study is based.
Gender-differences in learning outcomes | evaluation within 4 weeks after study completion
  Expert-based assessment of the difference in time (seconds) to the predefined primary critical action between randomized groups in video recordings of an in-person assessment simulation based on gender.
Group difference in global cognitive load while performing the in-person assessment simulation | evaluation within 4 weeks after study completion
  Assessment of the difference in global cognitive load between randomized groups immediately following the in-person assessment simulation using the National Aeronautics and Space Administration (NASA) global task load index, which ranges from 0 to 100. Higher scores indicate greater cognitive load.
Group difference in cognitive load (per objective) while performing the in-person assessment simulation | evaluation within 4 weeks after study completion
  Assessment of the difference in cognitive load (per objective) between randomized groups immediately following the in-person assessment simulation using the National Aeronautics and Space Administration (NASA) task load index, which ranges from 0 to 100.
  Objectives are: (mental demand, physical demand, temporal demand, performance, effort, frustration). Higher scores indicate greater mental demand/higher physical demand/ higher temporal demand/worse performance/more effort/more frustration).
Gaze behavior during the in-person assessment simulation: dwell-time in areas of interest | evaluation within 4 weeks after study completion
  Assessment of differences (in seconds) in gaze behavior (dwell time in areas of interest) using Tobii Pro eye-tracking technology between randomized groups based on recordings of the in-person assessment simulation
  The defined areas of interest for analysis are the manikin's head/airway, the manikin's thorax, the vital signs monitor, and the ventilator monitor.
Gaze behavior during the in-person assessment simulation: fixation count in areas of interest | evaluation within 4 weeks after study completion
  Assessment of differences in gaze behavior (fixation count in areas of interest) using Tobii Pro eye-tracking technology between randomized groups based on recordings of the in-person assessment simulation.
  The defined areas of interest for analysis are the manikin's head/airway, the manikin's thorax, the vital signs monitor, and the ventilator monitor.
Gaze behavior during the in-person assessment simulation: average fixation duration in areas of interest | evaluation within 4 weeks after study completion
  Assessment of differences (in seconds) in gaze behavior (average fixation duration in areas of interest) using Tobii Pro eye-tracking technology between randomized groups based on recordings of the in-person assessment simulation
  The defined areas of interest for analysis are the manikin's head/airway, the manikin's thorax, the vital signs monitor, and the ventilator monitor.
Gaze behavior during the in-person assessment simulation: time when no area of interest is illustrated | evaluation within 4 weeks after study completion
  Assessment of differences (in seconds) in gaze behavior (time when no area of interest is illustrated) using Tobii Pro eye-tracking technology between randomized groups based on recordings of the in-person assessment simulation
  The defined areas of interst for analysis are the manikin's head/airway, the manikin's thorax, the vital signs monitor, and the ventilator monitor.
Participants' subjective impressions of their learning progress when using virtual reality/e-learning | evaluation within 4 weeks after study completion
  5-point Likert scale
  1 - not helpful at all; 2 - rather not helpful; 3 - neither helpful nor not helpful; 4 - rather helpful; 5 - very helpful
Participants' subjective impressions of their level of frustration when using virtual reality/e-learning | evaluation within 4 weeks after study completion
  5-point Likert scale
  1 - not frustrated at all; 2 - rather not frustrated; 3 - neither frustrated nor not frustrated; 4 - rather frustrated; 5 - very frustrated
Participants' subjective impression of their level of enjoyment when using virtual reality/e-learning | evaluation within 4 weeks after study completion
  5-point Likert scale
  1 - not enjoyed at all; 2 - rather not enjoyed; 3 - neither enjoyed nor not enjoyed; 4 - rather enjoyed; 5 - very enjoyed
Participants' subjective confidence in recognizing and providing initial care to polytraumatized patients in cardiac arrest in the in-person assessment simulation | evaluation within 4 weeks after study completion
  5-point Likert scale
  1 - not confident at all; 2 - rather not confident; 3 - neither confident nor not confident; 4 - rather confident; 5 - very confident
Participants' subjective overall performance in the simulation sessions | evaluation within 4 weeks after study completion
  5-point Likert scale
  1 - not good at all; 2 - rather not good; 3 - neither good nor not good; 4 - rather good; 5 - very good
Participants' overall performance in the simulation sessions from the expert's point of view | evaluation within 4 weeks after study completion
  5-point Likert scale
  1 - not good at all; 2 - rather not good; 3 - neither good nor not good; 4 - rather good; 5 - very good
The correlation between how often participants have played virtual reality video games in the past 12 months and the primary outcome | evaluation within 4 weeks after study completion
  Spearman correlation
  Frequency of playing within the past 12 months: never; less than once a week; once per week; more than once per week; daily
The correlation between how often participants have played virtual reality video games between the ages of 6 and 18 and the primary outcome | evaluation within 4 weeks after study completion
  Spearman correlation
  Frequency of playing at the age of 6 to 18: never; less than once a week; once per week; more than once per week; daily
The correlation between how often participants have played non-virtual-reality video games in the past 12 months and the primary outcome | evaluation within 4 weeks after study completion
  Spearman correlation
  Frequency of playing within the past 12 months: never; less than once a week; once per week; more than once per week; daily
The correlation between how often participants have played non-virtual-reality video games between the ages of 6 and 18 and the primary outcome | evaluation within 4 weeks after study completion
  Spearman correlation
  Frequency of playing at the age of 6 to 18: never; less than once a week; once per week; more than once per week; daily
Incidence rate of virtual reality related adverse events | evaluation within 4 weeks after study completion
  Incidence of nausea, vomiting, dizziness, headache, overexertion/fatigue of the eyes (discomfort, blurred vision), stumbling, falling, bumping into real world objects while using virtual reality
System usability score for use of VR simulations | evaluation within 4 weeks after study completion
  System Usability Scale score from 1 to 100 points
Adjective Rating Scale for the use of the virtual reality simulations | evaluation within 4 weeks after study completion
  7-point Likert scale
  1 - the worst thing you can imagine; 2 - terrible; 3 - poor; 4 - okay; 5 - good; 6 - excellent; 7 - the best thing you can imagine

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lintschinger JM, Metelka P, Kapral L, Kahlfuss F, Reischmann L, Kaider A, Holaubek C, Kaiser G, Wagner M, Ettl F, Sixt L, Schaden E, Hafner C. Enhancing trauma cardiopulmonary resuscitation simulation training with the use of virtual reality (Trauma SimVR): Protocol for a randomized controlled trial. PLoS One. 2025 Jan 24;20(1):e0316828. doi: 10.1371/journal.pone.0316828. eCollection 2025. PMID 39854477